CLINICAL TRIAL: NCT00828867
Title: A Double-Blind, Parallel, Randomized, Placebo-Controlled, Single Dose Escalation First Time in Human Study to Investigate the Safety, Tolerability and Pharmacokinetics of Investigational Study Drug in Healthy Subjects
Brief Title: Single Dose Escalation First Time in Human PK Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 111341
Record Dates: First submitted 2008-12-08; First posted 2009-01-26 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Infections, Bacterial
Keywords: healthy subjects; FTIH, single dose, food effect, healthy subjects, double-blind
MeSH Terms: conditions — Bacterial Infections | interventions — Drug Evaluation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- Cohort 1 (Experimental): 100mg
  Interventions: Drug: 100 mg GSK investigational drug
- Cohort 2 (Experimental): 200mg
  Interventions: Drug: 200 mg GSK investigational drug
- Cohort 3 (Experimental): 400mg
  Interventions: Drug: 400 mg GSK investigational drug
- Cohort 4 (Experimental): 800mg
  Interventions: Drug: 800 mg GSK investigational drug
- Cohort 5 (Experimental): 1500mg
  Interventions: Drug: 1500 mg GSK investigational drug
- Cohort 6 (Experimental): 2000mg
  Interventions: Drug: 2000 mg GSK investigational drug
- Cohort 7 (Experimental): 800mg with food
  Interventions: Drug: 800mg fed GSK investigational drug
- Cohort 8 (Experimental): 3000mg
  Interventions: Drug: 3000mg GSK investigational drug
- Cohort 9 (Experimental): 4000mg
  Interventions: Drug: 4000mg GSK investigational drug

INTERVENTIONS:
Drug: 100 mg GSK investigational drug
  Other Names: selected mg fed study drug; 2000 mg study drug; 800 mg study drug; 400 mg study drug; 200 mg study drug; 100 mg study drug; 1500 mg study drug
  Arms: Cohort 1
Drug: 200 mg GSK investigational drug
  Arms: Cohort 2
Drug: 400 mg GSK investigational drug
  Arms: Cohort 3
Drug: 800 mg GSK investigational drug
  Arms: Cohort 4
Drug: 2000 mg GSK investigational drug
  Arms: Cohort 6
Drug: 1500 mg GSK investigational drug
  Arms: Cohort 5
Drug: 800mg fed GSK investigational drug
  Arms: Cohort 7
Drug: 3000mg GSK investigational drug
  Arms: Cohort 8
Drug: 4000mg GSK investigational drug
  Arms: Cohort 9

SUMMARY:
This is a first time in human (FTIH) study of single escalating doses of investigational study drug to investigate safety, tolerability, and pharmacokinetics in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* male
* non-childbearling potential females
* Body weight greater than or equal to 50 kg (110 lbs) for men and greater than or equal to 45 kg (99 lbs) for women. Body mass index (BMI) between 18.5-29.9 kg/m2 inclusive.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* QTcB < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block on Screening ECG

Exclusion Criteria:

* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as:

an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males), or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). A standard unit is defined as 10g ethanol which is equivalent to 100mL wine, 250mL full strength beer, 470mL light beer, 30mL spirits

* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive [serum or urine] human chorionic gonadotropin (hCG) test at screening or prior to dosing.
* Lactating females.
* Subjects who have asthma or a history of asthma within the past 6 months.
* History of smoking or history of regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice, pummelos, satsuma, ugli, tangerine, and tangelo, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-11-14 (Actual); Primary Completion 2009-12-07 (Actual); Study Completion 2009-12-07 (Actual)

PRIMARY OUTCOMES:
Safety parameters, adverse events, absolute values and changes over time of hematology, clinical chemistry, urinalysis, vital signs, electrocardiogram intervals, and ECG rhythm. | Eighteen days
Pharmacokinetic parameters following single dose administration: area under the plasma concentration curve AUC 0 to inf, AUC 0 to t, AUC 0 to 24, maximum observed concentration , time to maximum observed concentration , terminal half life . | Two days, Three days (3000mg and 4000mg only)

SECONDARY OUTCOMES:
AUC 0 to inf and Cmax following single dose administration for the assessment of dose proportionality | Two days, Three days (3000mg and 4000mg only)
Amount excreted of unchanged study drug and renal clearance | Two days, Three days (3000mg and 4000mg only)
AUC 0 to inf, AUC 0 to t, AUC 0 to 24, Cmax, tmax and tlag if deemed appropriate with and without high fat calorie meal | Two days, Three days (3000mg and 4000mg only)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Naderer OJ, Dumont E, Zhu J, Kurtinecz M, Jones LS. Single-dose safety, tolerability, and pharmacokinetics of the antibiotic GSK1322322, a novel peptide deformylase inhibitor. Antimicrob Agents Chemother. 2013 May;57(5):2005-9. doi: 10.1128/AAC.01779-12. Epub 2013 Feb 12. PMID 23403431
- See also: Results for study 111341 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/111341?search=study&search_terms=111341#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 111341 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111341 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111341 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111341 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111341 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111341 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111341 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register